CLINICAL TRIAL: NCT00614354
Title: Phase II Study of 99mTc-glucarate in Chest Pain Patients Suspected With ACS With no Obvious Signs of AMI and With Known Previous CAD.
Brief Title: Study of 99mTc-glucarate to Detect Acute Coronary Syndrome in Chest Pain Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Molecular Targeting Technologies, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Yale University (Other); University of Pittsburgh (Other); University of Alabama at Birmingham (Other); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MTTI ACS 201; 5R44HL062770-06 (NIH)
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Acute Coronary Syndrome
Keywords: 99mTc-glucarate imaging to detect acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: 99mTc-glucarate solution

INTERVENTIONS:
Drug: 99mTc-glucarate solution — Patients will receive a single 22 - 27 mCi bolus intravenous dose of 99mTc-glucarate solution, as soon as possible after their arrival in the emergency department or the chest pain center

SUMMARY:
The purpose of this clinical trial is to study the ability of a radioactive drug called "Technetium Glucarate" to detect whether the cause of chest pain in patients entering the emergency department with no obvious signs of heart attack is due to a condition called Acute Coronary Syndrome (ACS). The drug will be injected intravenously. After one or two hours the patient will undergo an imaging procedure to detect if the drug has accumulated in the heart. Uptake of the radioactive drug in the heart is indicative of reduced blood flow to the heart.

DETAILED DESCRIPTION:
Acute coronary syndrome encompasses a range of coronary artery diseases, including unstable angina and both ST-segment elevation and non-ST-segment elevation myocardial infarction (MI). Differentiating ACS from noncardiac chest pain remains a challenge in the emergency department (ED). Myocardial perfusion imaging (MPI) for ischemia has been used to rule ACS in or out among chest pain patients with nondiagnostic ECGs upon presentation to the ED. Several studies have shown a high negative predictive value of MPI for ruling out acute ischemia in the emergency setting. Although myocardial imaging with perfusion agents provides important information for risk-stratifying stable post-ACS patients, this method is of limited value in patients with prior history of CAD, since these patients will often have abnormal resting perfusion patterns, thereby precluding the ability to differentiate old infarcts from new ischemic events. 99mTc-glucarate does not detect old MIs and thus should provide an improvement in specificity in the imaging of ACS patients with previous CAD.

This study proposes to extend the evaluation of 99mTc-glucarate imaging by studying its ability to detect ACS in chest pain patients with no obvious signs of AMI but with known CAD, in the setting of the ED. Unlike MPI, 99mTc-glucarate imaging will not detect old MIs, thereby providing an advantage in specificity of the technique.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain of recent onset (less than 24 hours) and of greater than 5-minute duration, consistent with ACS;
* History of CAD;
* Creatinine level less than 3.5 mg per deciliter;
* Female patients who are: surgically sterile (hysterectomy or bilateral tubule libation), at least one year post-menopausal, or have a negative pregnancy test on the day of treatment; and
* Written informed consent.
* This research is being supported by the NIH/NHLBI which requires a minimum 50% participation from women. Efforts should be made to enroll equal numbers of men and women at each clinical site.

Exclusion Criteria:

* ECG changes diagnostic of AMI;
* A cardiac revascularization procedure within the last 2 weeks (non-revascularization procedures such as cardiac catheterization, stress test or echocardiography are acceptable);
* An alternate diagnosis more probable than ACS;
* Presence of pericarditis, myocarditis, acute aortic dissection, pneumothorax, or pulmonary embolism (PE);
* Patients with uncontrolled severe heart failure at the time of enrollment (NYHA class III and IV).
* Other serious or life-threatening disease that might preclude a subject from completing this study;
* Clinically essential procedures with which this protocol may interfere;
* Previous 99mTc-based diagnostic test within the last 24 hours;
* Female subjects who are pregnant or lactating;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Readers will assess images as either positive or negative and note the location of uptake. | Immediately and end of enrolement

CONTACTS AND LOCATIONS:
Overall Officials: Albert J. Sinusas, MD, Principal Investigator — Yale University; Diwakar Jain, MD, Study Chair — Drexel University; Prem Soman, MD, Ph.D., Principal Investigator — University of Pittsburgh; Ami E Iskandrian, MD, Principal Investigator — University of Alabama at Birmingham; Robert S Jones, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Yale University, New Haven, Connecticut
  - University Hospital Case Medical Center, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania